CLINICAL TRIAL: NCT06640608
Title: Efficacy of Internet- Based Cognitive Behavioral Therapy Among Women With Fear of Childbirth: A Randomized Controlled Trial
Brief Title: Internet- Based Cognitive Behavioral Therapy Among Women With Fear of Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jouf University (Other)
Responsible Party: Principal Investigator, Enas Mahrous AbdelAziz, Assistant professor of psychiatric mental health nursing, Jouf University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 64
Record Dates: First submitted 2024-10-05; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Pregnant Women; Fear of Childbirth; Self Efficacy; Cognitive Behavioral Therapy
Keywords: pregnant women; Fear of Childbirth; Self Efficacy; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: the study compare between intervention group (internet -based cognitive behavioral therapy therapy in addition to stander of care and the usual stander of care
Who Masked: Participant, Outcomes Assessor
Masking Description: Study participants and Outcome assessors are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group ( received ICBT in addition to routine antenatal care) (Experimental): provide 6 consecutive an online modules
  Interventions: Behavioral: ICBT - Internet Based Cognitive Behavioral Therapy
- Control group (No Intervention): Received routine antenatal care only

INTERVENTIONS:
Behavioral: ICBT - Internet Based Cognitive Behavioral Therapy — The study (intervention) group received 6 consecutive sessions utilizing ICBT techniques to overcome Fear of childbirth
  Arms: intervention group ( received ICBT in addition to routine antenatal care)

SUMMARY:
Fear of Birth is common in pregnant women and associated with physiological and psychological consequences. Fear is mostly associated with fear of losing control, fear for the baby's life or health or own life threatening events .

Cognitive Behaviour Therapy (CBT) is the treatment of choice for most anxiety disorders and for women with mental health problems during pregnancy and postpartum.. It has been suggested for perinatal women as with Fear of Birth. Internet-based cognitive behavioural therapy have shown it is efficiency as treatment for anxiety and depression as traditional face-to-face CBT in managing emotional problems for women

DETAILED DESCRIPTION:
Fear of Birth is common in pregnant women , the current study aims to examine the efficacy of an Internet-based Cognitive behavioral therapy compared to standard of care for women with fear of child birth( moderate /severe).

The study comparing internet -based Cognitive Behavioral therapy in addition to routine stander of antenatal care (interventional group) with others who are receiving stander of care alone( control group). The study is the second phase of the study project named "Prevalence of childbirth fear and associated factors among pregnant women.

based on inclusion and exclusion criteria, the total participants who have moderate and severe level of child birth fear is 169 pregnant women . The final sample eligible is 96 participants . Those will assign randomly to either interventional / control group

the interventional group will receive internet -based cognitive behavioural therapy program accompanied with stander of care providing at antenatal clinics . through whats app group the researchers will provide the program contents

ELIGIBILITY:
Inclusion Criteria:

* accepting and willing to engage in an ICBT program
* participants experienced a fear of childbirth score ranging from 40 to 64 based on the Childbirth Attitude Questionnaire (CAQ)
* Aged between 18 and 35 years
* Gestational age of at least 28 weeks (determined by an accurate last menstrual period)
* singleton pregnancy
* (Capability to read, write, and understand the essence of the provided questionnaires
* have a smartphone with internet access
* had not participated in any antenatal intervention or education.

Exclusion Criteria:

* women diagnosed with pathological anxiety or depression
* Pregnancies associated with serious health issues (e.g., hypertension, infections, diabetes, obesity, etc.)
* A recent history of pregnancy complications
* women not respond for at least two modules of intervention program
* A recent history of miscarriage or neonatal loss
* A history of infertility
* Lack of access to the internet.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female only
Enrollment: 96 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Change Childbirth fears | 6 weeks intervention
  Pregnant women who receive an internet -based Cognitive Behavioral Therapy education report a significant change in a mean scores of fear of childbirth than those in a control group.
  Childbirth Attitude Questionnaire (CAQ) was used to assess childbirth fear. Scores range from 16 to 64, with higher scores indicating greater fear of childbirth. The CAQ categorizes scores into four levels: low (16-27), mild (28-39), moderate (40-51), and severe (52-64).
Increase self-efficacy | 6 weeks intervention
  Pregnant women who receive an internet-based Cognitive Behavioral Therapy education report a significant change in mean scores of maternal self-efficacy than those in a control group.
  The Childbirth Self- Efficacy Inventory (CBSEI) was used including 32 items separating it into two distinct stages. The scale includes two parallel subscales: the outcome expectancy subscale measures the belief that certain behaviors will lead to specific outcomes, while the efficacy expectancy subscale assesses confidence in one's ability to perform these behaviors. Both subscales consist of the same 16 items related to coping behaviors during childbirth. Responses are rated on a Likert scale from 1 to 10, with higher scores reflecting greater self-efficacy in childbirth.

CONTACTS AND LOCATIONS:
Locations (1):
- Governmental Clinics, Beheira, Egypt

REFERENCES:
- [Derived] Abdelaziz EM, Alshammari AM, Elsharkawy NB, Oraby FA, Ramadan OME. Digital intervention for tokophobia: a randomized controlled trial of internet-based cognitive behavioral therapy on fear of childbirth and self-efficacy among Egyptian pregnant women. BMC Pregnancy Childbirth. 2025 Mar 3;25(1):233. doi: 10.1186/s12884-025-07341-5. PMID 40033245